CLINICAL TRIAL: NCT01854853
Title: Brazilian HIV/Sexually Transmitted Infection (STI) Prevention for Adolescents With Mental Health
Brief Title: Brazilian HIV/Sexually Transmitted Infection (STI) Prevention for Adolescents With Mental Health Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 6394; R34MH094163 (NIH)
Record Dates: First submitted 2013-05-02; First posted 2013-05-16 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: HIV; Sexually Transmitted Infection; Pregnancy
Keywords: unsafe sex; safer sex; HIV; STI; Pregnancy
MeSH Terms: conditions — Sexually Transmitted Diseases; Unsafe Sex | interventions — Health Promotion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STYLE Brazil (Experimental): STYLE-BRazil Multifamily Group HIV/STI Prevention intervention
  Interventions: Behavioral: STYLE Brazil
- Health Promotion (Active Comparator): Health Promotion Intervention - Adolescents only
  Interventions: Behavioral: Health Promotion

INTERVENTIONS:
Behavioral: STYLE Brazil — Multifamily group HIV/STI Prevention Intervention
  Arms: STYLE Brazil
Behavioral: Health Promotion — Health promotion intervention
  Arms: Health Promotion

SUMMARY:
Adolescents with mental health (MH) disorders (MHD) have higher rates of HIV/STI sexual risk behaviors than those in the general population. In Brazil, among youth seeking HIV testing, those testing positive had more MH problems than HIV-negative youth; HIV/STI sexual risk reduction is not regularly implemented within MH care for adolescents. Our NIMH-funded RCT in Rio de Janeiro (Rio; R01MH065163; PI: Wainberg) promises to provide such intervention for adults with MHD. A comparable evidence-based HIV/STI prevention intervention for adolescents is not available in Brazil; this application targets this need.

Using quantitative and qualitative methods we will explore the contextual influences on sexual risk behavior of Brazilian youth ages 13-24 with MHD to inform intervention adaptation. The investigators will then pilot-test the family-based (parent-adolescent dyad) intervention HIV, STI and pregnancy prevention intervention with a sample of male and female youth age 13-24 years (n=144) with MHD who are in MH treatment in four community-based sites in preparation for the RCT.

DETAILED DESCRIPTION:
Adolescents with mental health (MH) disorders (MHD) have higher rates of HIV/STI sexual risk behaviors than those in the general population. In Brazil, among youth seeking HIV testing, those testing positive had more MH problems than HIV-negative youth; HIV/STI sexual risk reduction is not regularly implemented within MH care for adolescents. Our NIMH-funded RCT in Rio de Janeiro (Rio; R01MH065163; PI: Wainberg) promises to provide such intervention for adults with MHD. A comparable evidence-based HIV/STI prevention intervention for adolescents is not available in Brazil; this application targets this need. To address this public health need and opportunity, we propose to a) adapt a U.S. efficacious family-based HIV prevention intervention for youth with MHD (STYLE; R01MH63008; PI: Brown) within the three types of settings providing most of the care to adolescents with MHD in Brazil; and b) pilot test the intervention to examine the acceptability, feasibility, and implementation parameters of the resulting Brazil intervention (STYLE-B) within these settings, and to determine key research parameters in preparation for an implementation randomized clinical trial (RCT). Using quantitative and qualitative methods we will explore the contextual influences on sexual risk behavior of Brazilian youth ages 13-24 with MHD to inform intervention adaptation. The investigators will then pilot-test STYLE-B with a sample of male and female youth age 13-24 years (n=144) with MHD who are in MH treatment in four community-based sites. Youth/caregiver dyads will receive a full-day group session, return in two weeks for an adolescent/caregiver dyad session, and participate in a half-day group session three months later. Acceptability and feasibility will be assessed using process measures after each session. The investigators will assess change in sexual risk behavior outcomes from baseline to 3-months post-intervention. The investigators will elucidate factors influencing intervention adoption (e.g., recruitment, referrals; resources; climate, readiness and capacity for intervention) within the three service systems for youth with MHD in Brazil. The investigators will develop digital web-based interactive technology to train intervention facilitators in preparation for the RCT.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent with a mental health disorder in any of the four pilot sites;
* Ages 13-24;
* having a caregiver who is willing to participate and sign consent for their adolescent's involvement in the study.

Exclusion Criteria:

* primary alcohol or other drug use disorder (AOD);
* mental retardation or pervasive developmental disorder as primary diagnosis;
* a medical or psychiatric illness requiring hospitalization; and
* currently psychotic or suicidal.

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 305 (Actual)
Dates: Start 2012-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
AIDS Risk Behavior Assessment (ARBA) | In the past 3 months
  We will assess sexual activity, unprotected sex acts and number of sexual partners (if sexually active) or delay sexual debut (if not sexually active) in the last 3 months at baseline and 3 months post intervention

SECONDARY OUTCOMES:
Parent-adolescent communication about sex scale | Past 3 months
  The measure assess parent adolescent communication about sex in the last 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Milton L Wainberg, MD, Principal Investigator — NYSPI/Columbia University
Locations (1):
- CAPSi João Caetano, Itaboraí, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Wainberg ML, McKinnon K, Mattos PE, Pinto D, Mann CG, de Oliveira CS, de Oliveira SB, Remien RH, Elkington KS, Cournos F; PRISSMA Project. A model for adapting evidence-based behavioral interventions to a new culture: HIV prevention for psychiatric patients in Rio de Janeiro, Brazil. AIDS Behav. 2007 Nov;11(6):872-83. doi: 10.1007/s10461-006-9181-8. Epub 2007 Jan 10. PMID 17216334